CLINICAL TRIAL: NCT03480529
Title: Monitoring the IMmUological TOXicity of Drugs
Acronym: MIMUTOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Joe Elie Salem, MD,PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-05
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Arthritis; Systemic Lupus Erythematosus; Rheumatoid Arthritis; Capillary Leak Syndrome; Hepatitis
Keywords: adverse event; arthritis; Systemic Lupus Erythematosus; Capillary Leak Syndrome; Hepatitis
MeSH Terms: conditions — Arthritis; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Capillary Leak Syndrome; Hepatitis | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Arthritis or lupus or CLS induced by a drug: Case reported in the World Health Organization (WHO) of arthritis or lupus, or Hepatitis, or capillary leak syndrome of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: drug inducing arthritis, lupus, hepatitis, or capillary leak syndrom

INTERVENTIONS:
Drug: drug inducing arthritis, lupus, hepatitis, or capillary leak syndrom — Drugs susceptible to induce arthritis, lupus, hepatitis, or capillary leak syndrom

SUMMARY:
Several drugs and chemotherapies seem to have an impact on the immunological system. This study investigates reports of immunological toxicities, including the International classification of disease ICD-10 codes M05, M32, I78 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the immunological system and are responsible of a wide range of rare immunological side effects. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by rare immunological side effects (of which systemic lupus, immune arthritis, rheumatoid arthritis, Hepatitis, capillary leak syndrome) imputed to drugs. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 02/01/2018
* Adverse event reported were including the MedDRA terms for immune arthritis, systemic lupus erythematosus, hepatitis, rheumatoid arthritis and capillary leak syndrome.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Arthritis, hepatitis, and lupus induced toxicity of Immune Checkpoint inhibitors (ICI) Identification and report of cases of arthritis or lupus associated with ICIs. The research includes the report with MedDRA terms: | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018

SECONDARY OUTCOMES:
Causality assessment of reported arthritis, hepatitis, or lupus events according to the WHO system | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the type of arthritis or lupus or hepatitis or capillary leak syndrom depending on the category of drug | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the other immune related adverse events concomitant to the arthritis or lupus or hepatitis or capillary leak syndrom induced by drugs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018
Description of the population of patients having a arthritis or lupus or hepatitis or CLS adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 02/01/2018

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris
  - Rhumatology department, CHU Strasbourg, Hautepierre hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnaud L, Lebrun-Vignes B, Salem JE. Checkpoint inhibitor-associated immune arthritis. Ann Rheum Dis. 2019 Jul;78(7):e68. doi: 10.1136/annrheumdis-2018-213470. Epub 2018 May 3. No abstract available. PMID 29724725
- [Result] Mertz P, Lebrun-Vignes B, Salem JE, Arnaud L. Characterizing drug-induced capillary leak syndromes using the World Health Organization VigiBase. J Allergy Clin Immunol. 2019 Jan;143(1):433-436. doi: 10.1016/j.jaci.2018.09.001. Epub 2018 Sep 20. No abstract available. PMID 30244023
- [Result] Arnaud L, Mertz P, Gavand PE, Martin T, Chasset F, Tebacher-Alt M, Lambert A, Muller C, Sibilia J, Lebrun-Vignes B, Salem JE. Drug-induced systemic lupus: revisiting the ever-changing spectrum of the disease using the WHO pharmacovigilance database. Ann Rheum Dis. 2019 Apr;78(4):504-508. doi: 10.1136/annrheumdis-2018-214598. Epub 2019 Feb 4. PMID 30793701